CLINICAL TRIAL: NCT04490902
Title: Suppression of Graft Rejection Using Mixed Component Cornea in the High-risk Keratoplasty，A Randomized Controlled Trial.
Brief Title: Clinical Study on the Treatment of Mixed Component Cornea for High Risk Keratoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020KYPJ111
Record Dates: First submitted 2020-07-22; First posted 2020-07-29 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Corneal Transplantation
Keywords: High-risk corneal transplantation; Penetrating keratoplasty; Limbal transplantation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single graft corneal transplantation (Active Comparator): Limbal transplantation combined with central penetrating keratoplasty from single donors.
  Interventions: Procedure: Limbal transplantation combined with central penetrating keratoplasty
- Dual graft corneal transplantation (Experimental): Limbal transplantation combined with central penetrating keratoplasty from different donors.
  Interventions: Procedure: Limbal transplantation combined with central penetrating keratoplasty

INTERVENTIONS:
Procedure: Limbal transplantation combined with central penetrating keratoplasty — Limbal transplantation combined with central penetrating keratoplasty with single donor cornea
  Arms: Single graft corneal transplantation
Procedure: Limbal transplantation combined with central penetrating keratoplasty — Limbal transplantation combined with central penetrating keratoplasty with mixed component cornea
  Arms: Dual graft corneal transplantation

SUMMARY:
Because of the immunologically privileged nature of the cornea, the graft rejection rate is less than 10% for low-risk keratoplasty. But when the cornea performed 2 or more quadrants of corneal neovascularization after ocular trauma or infection, the graft rejection rate is more than 65%, it is called high-risk keratoplasty.

This study will observe the graft survival of high-risk corneal transplantation using mixed component cornea from different donors.

DETAILED DESCRIPTION:
Ocular trauma or infection lead to corneal limbal stem cell deficiency and central corneal opacification which could only be treated by central penetrating keratoplasty and limbal transplantation, but the rejection rate is very high. In clinical, we found that limbal transplantation combined with central penetrating keratoplasty from different donors can keep the graft transparent for a long time, this result also be found in organ transplantation, multiple donor organ transplantation could reduce rejection risk in liver and kidney transplantation. Therefore, it is speculated that there are different MHC antigens from different donors, which cause different reactions after transplantation. Because there are a large number of Langerhans cells， abundant blood vessels and lymphatic in the limbal, so the rejection occurs early and severely. Continuous and intense limbal rejection leads to the depletion of recipient T cells, lead to the immune tolerance of another donor's central corneal tissue. In this project, central penetrating keratoplasty and limbal transplantation from different donors will be carried out and the graft survival of high-risk corneal transplantation will be observed in clinical, to find a new method for high-risk corneal transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Central corneal opacity involving full layer
* Corneal neovascularization in two or more quadrants
* Patients must be willing and able to return for scheduled follow-up examinations for 12 months after surgery
* Ages：18 -70 Years

Exclusion Criteria:

* Central corneal opacity not involving the endothelial layer
* Less than two quadrants of corneal neovascularization
* History of Stevens-Johnson syndrome or Sjogren's syndrome
* Severe eyelid and conjunctival scar
* Loss of vision in contralateral eye
* Pregnant and lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-08-18 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
The rate of corneal graft rejection at 12 months | 12 months
  The rejection index of corneal transplantation will be observed by slit lamp after surgery

SECONDARY OUTCOMES:
The changes of best corrected visual acuity | Before surgery, 1 week, 1 month, 3 months, 6 months, 12 months
  Best corrected visual acuity in different point will be compared with preoperative
The changes of corneal thickness depth | baseline (Before surgery), 1 week, 1 month, 3 months, 6 months, 12 months
  Corneal thickness depth will be measured by anterior segmental OCT and compared with preoperative
Reconstruction of corneal limbal | baseline (Before surgery), 1 week, 1 month, 3 months, 6 months, 12 months
  Confocal microscopy will be used to define whether the structure of corneal limbal has reconstructed
Endothelial Cell Density | baseline (Before surgery), 1 week, 1 month, 3 months, 6 months, 12 months
  Endothelial Cell Density will be measured by specular microscope to evaluate the loss of endothelial cells
The rate of presence of goblet cells containing conjunctival epithelium on the corneal surface by impression cytology | baseline (Before surgery), 1 week, 1 month, 3 months, 6 months, 12 months
  Detects whether conjunctival epithelial and goblet cells have invaded the corneal surface by impression cytology, to observe the reconstruction of limbal function

OTHER OUTCOMES:
Intraocular pressure | Before surgery, 1 week, 1 month, 3 months, 6 months, 12 months
  Intraocular pressure will be measured by non contact tonometer as safety index

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No